CLINICAL TRIAL: NCT04099836
Title: Single Arm Phase 2 Trial of Atezolizumab and Bevacizumab in Epidermal Growth Factor Receptor (EGFR) Mutant Non-Small Cell Lung Cancer in Patients With Progressive Disease After Receiving Osimertinib (TOP 1901)
Brief Title: Atezolizumab and Bevacizumab in EGFR Mutant NSCLC in Patients With Progressive Disease After Receiving Osimertinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103723
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR Mutation; Atezolizumab; Bevacizumab; exon L858R; exon 21 L858R
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- atezolizumab and bevacizumab (Experimental): Atezolizumab 1200 mg IV every 3 weeks and bevacizumab 15 mg/kg IV every 3 weeks (1 cycle=3 weeks)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV every 3 weeks
  Other Names: TECENTRI
Drug: Bevacizumab — 15 mg/kg IV every 3 weeks
  Other Names: Avastin

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of giving atezolizumab combined with bevacizumab in patients with stage 4 epidermal growth factor receptor (EGFR) mutant non-small cell lung cancer (NSCLC) whose cancer has gotten worse while receiving osimertinib.

DETAILED DESCRIPTION:
This study will be single arm, open label, phase 2 study which will include patients with stage 4 NSCLC patients with EGFR mutations and who have progressed on osimertinib.

Although both atezolizumab and bevacizumab are approved for the treatment of NSCLC, the combination of atezolizumab and bevacizumab has not been approved by the FDA for the treatment of specific non-small cell lung cancer (NSCLC).

Patients who have one of the following EGRF mutations: exon 19 or exon 21 L858R with progressive disease on osimertinib may be eligible to participate in this study. If enrolled into the study, the study team will give the patient atezolizumab (1200 mg) combined with bevacizumab (15 mg/kg) every 3 weeks intravenously. As part of this study, the patient will have blood samples, other tests, exams, and procedures done for study purposes and their standard of care. Patient participation in the study will last for up to 2 years after completion of the last dose of the study drug or until your condition worsens or intolerable adverse events as deemed by the study doctor.

There are possible patient risks to this study that include but are not limited to diarrhea, itching, rash, and a feeling of weakness.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologic documentation of primary lung carcinoma, non-squamous histology with EGFR exon deletion 19 or exon 21 L858R mutation
3. Stage IV disease according to the 8th Edition of the American Joint Committee on Cancer staging system
4. Disease progression on osimertinib
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 (appendix 1)
6. Measureable disease as defined by RECIST 1.1 (appendix 2)
7. The following laboratory values obtained ≤ 30 days prior to starting study therapy

   1. ANC ≥ 1, 500 / mm3
   2. Platelet count, ≥ 100,000 / mm3
   3. Hemoglobin ≥ 9.0 g / dL
   4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   5. Serum Glutamic Oxaloacetic Transaminase (SGOT) (Aspartate Aminotransferase, AST) and Serum Glutamic Pyruvic Transaminase (SGPT) (Alanine Aminotransferase, ALT) ≤2.5 x ULN in patients without liver or bone metastases; < 5 x ULN in patients with liver or bone metastases.
   6. Cockcroft-Gault calculated creatinine clearance of ≥ 45 ml/min (appendix 3) or creatinine ≤1.5 x ULN
   7. Urine protein/creatinine (UPC) ratio ≤1.
8. Negative pregnancy test done ≤7 days (or per institutional policy) prior to start of study therapy, for women of childbearing potential only. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test of must have evidence of non-child bearing potential by fulfilling one of the following criteria at screening:

   1. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments;
   2. Women under 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and Luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution;
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
9. Male subjects should be willing to use barrier contraception.
10. Provide informed written consent

Exclusion Criteria:

1. Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component.
2. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown: pregnant women, nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception
3. Other active malignancy ≤ 2 years prior to study cycle 1 day 1 of study therapy. EXCEPTIONS: Nonmelanotic skin cancer or carcinoma-in-situ of the cervix, or adequately treated stage I or II cancer. NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (i.e. hormonal therapy) for their cancer.
4. History of myocardial infarction or other evidence of arterial thrombotic disease (angina), symptomatic congestive heart failure (New York Heart Association ≥ grade 2), unstable angina pectoris, or ventricular arrhythmia with ≤ 6 months
5. History of cerebral vascular accident (CVA) or transient ischemic attack (TIA) ≤ 6 months prior to study cycle 1 day 1 of study therapy.
6. History of bleeding diathesis or coagulopathy.
7. Inadequately controlled hypertension (systolic blood pressure of >160 mmHg or diastolic pressure >100 mmHg on anti-hypertensive medications). Note: History of hypertensive crisis or hypertensive encephalopathy not allowed.
8. Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury ≤ 28 days or core biopsy ≤ 7 days prior to starting therapy
9. History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess ≤6 months prior to study cycle 1 day 1 of study therapy.
10. Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
11. History of hemoptysis ≥ grade 2 (defined as bright red blood of at least 2.5 mL) ≤ 3 months prior to cycle 1 day 1 of study therapy.
12. Symptomatic untreated brain metastases which is defined as persistent neurological symptoms or requiring ongoing use of steroids. Asymptomatic untreated brain metastases are allowed if ≤ 1 cm
13. Significant vascular disease (e.g. aortic aneurysm surgical repair or recent peripheral arterial thrombosis) ≤6 months prior to starting study therapy
14. Radiotherapy to any site for any reason ≤ 14 days prior to study cycle 1 day 1 of study therapy.
15. Pre-existing and clinically active interstitial lung disease
16. Autoimmune condition requiring ongoing or intermittent systemic treatment. Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study treatment initiation. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

    Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
17. Prior therapy with anti-PD-1 or anti-PD-L1 immunotherapy,
18. Prisoners, participants who are involuntarily incarcerated, or participants who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant level data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab and Bevacizumab: Atezolizumab 1200 mg IV every 3 weeks and bevacizumab 15 mg/kg IV every 3 weeks (1 cycle=3 weeks)
  Atezolizumab: 1200 mg IV
  Bevacizumab: 15 mg/kg IV
Period: Overall Study
Arm/Group | Atezolizumab and Bevacizumab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab and Bevacizumab
Number analyzed (Participants) | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [61 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, cannot carry on any selfcare, totally confined to bed or chair; 5 = Dead
  Participants
    PS=0 | 7
    PS=1 | 0
    PS=2 | 0
    PS=3 | 0
    PS=4 | 0
    PS=5 | 0
EGFR mutation [Count of Participants; unit: Participants]
  Exon 19 | 3
  21 L858R | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Assessed by the Investigator Using RECIST 1.1
Description: Objective response (complete or partial response) rate (ORR) is assessed by the investigator using Response Evaluation Criteria in Solid Tumors RECIST 1.1 (brand name) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab and Bevacizumab
Number analyzed (Participants) | 7
Participants
  Overall response (OR) = CR + PR | 0
  Non-response (stable disease or progression) | 7

2. Secondary Outcome: Progression Free Survival as Measured by RECIST v1.1 RECIST 1.1 (Brand Name) as Assessed by the Investigator.
Description: Progression will be defined as time from start of study therapy to disease progression or death whichever comes first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median survival time and its 95% CI will be calculated.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab
Number analyzed (Participants) | 7
months | 2.1 [0.5 to NA] — The upper level of the 95% CI was not estimable at the time of analysis

3. Secondary Outcome: Overall Survival as Noted by Follow-up Via Composite of Telephone or Medical Record Review.
Description: Overall survival (OS) is defined as the time from start of study therapy to death from any cause, and patients who are alive at the time of analysis will be censored at the last date of contact.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab and Bevacizumab
Number analyzed (Participants) | 7
Months | 6.4 [3.2 to NA] — The upper level of the 95% CI was not estimable at the time of analysis

4. Secondary Outcome: Number of Participants With AEs as Measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: All patients who receive at least one dose of study treatment will be included in the safety analysis. The frequencies and percentage of treatment-related adverse events will be tabulated.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab and Bevacizumab
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Atezolizumab and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab and Bevacizumab (N=7)
Figure (General disorders) | 1
heart failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab and Bevacizumab (N=7)
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 2
Blurred vision (Eye disorders) | 2
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Ear and labyrinth disorders - intermittent ear fullness (Ear and labyrinth disorders) | 1
Eye disorder - loss peripheral vision bilaterally (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 4
Gastrointestinal disorders - Intermittent early satiety (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 2
Headache (Nervous system disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Memory impairment (Nervous system disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Intermittent loss in balance (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Investigations) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures - Pleurex right chest wall (Surgical and medical procedures) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary tract infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04099836/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT04099836/ICF_001.pdf